CLINICAL TRIAL: NCT01837446
Title: Evaluating the Effectiveness of Topical Morphine Compared With a Routine Mouthwash in Managing Cancer Treatment-induced Mucositis in Patients With Head and Neck Cancer in Isfahan
Brief Title: Morphine Mouthwash for Management of Oral Mucositis in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Simin Hemati, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 390163
Record Dates: First submitted 2013-02-26; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Stomatitis
Keywords: mucositis; topical morphine; pain; head and neck carcinoma
MeSH Terms: conditions — Stomatitis; Mucositis; Pain | interventions — aluminum hydroxide, magnesium hydroxide, drug combination; Lidocaine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine mouthwash (Experimental): The morphine group uses the mouthwash of 2% morphine solution (20 mg morphine sulfate diluted in 100 mL of water), 10 mL every three hours; six times a day. The morphine solution is prepared by the faculty of pharmacy under supervision of the Food and Drug Organization of the local Medical University.
  Interventions: Drug: 2% morphine solution
- Magic mouthwash (Active Comparator): The magic group uses a mouthwash contained a mixture of 240 mL magnesium aluminum hydroxide (Alborz Co., Iran), 25 mL 2% viscous lidocaine (SinaDaru Co., Iran), and 60 mL diphenhydramine (Emad Co., Iran), 10 mL every three hours; six times a day.
  Interventions: Drug: Magnesium aluminum hydroxide; Drug: 2% viscous lidocaine; Drug: Diphenhydramine

INTERVENTIONS:
Drug: 2% morphine solution
  Arms: Morphine mouthwash
Drug: Magnesium aluminum hydroxide
  Arms: Magic mouthwash
Drug: 2% viscous lidocaine
  Arms: Magic mouthwash
Drug: Diphenhydramine
  Arms: Magic mouthwash

SUMMARY:
Oral mucositis is a debilitating side effects of cancer treatment for which there is not much successful treatments at yet. The investigators are going to evaluate the effectiveness of topical morphine compared with a routine mouthwash in managing cancer treatment-induced mucositis. The investigators hypothesize that topical morphine is more effective and more satisfied by patients than the magic mouthwash in reducing severity of cancer treatment-induced oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients
* Severe oral mucositis; grade III or IV of the World Health Organization (WHO) rating of global mucositis
* Willingness to participate

Exclusion Criteria:

* History of severe renal or hepatic insufficiency
* Collagen-vascular disease
* Allergic reaction to morphine
* Current smokers or alcohol users
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mucositis severity | Up to six days
  Patients are visited by a radiation oncologist at baseline, 3rd day, and 6th day of the intervention. The WHO grading system of mucositis is administered for each patient in which, 0 indicates a healed mucositis and no signs or symptoms, 1 indicates mild soreness but not problem in eating, 2 indicates painful erythema, edema, or ulcers but able to eat, 3 indicates severe painful erythema, edema, or ulcers and having problem in eating, and 4 indicates if there is a requirement for parenteral or enteral support.

SECONDARY OUTCOMES:
Patient's satisfaction | After six days
  Patients also are asked about if pain/discomfort relived by mouthwash and if so for how long (< 1 h, 1 to 2 h, > 2 h). Their satisfaction with treatment is graded as satisfied, tolerable, and intolerable.

CONTACTS AND LOCATIONS:
Overall Officials: Simin Hemati, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Radiation Oncology Department, Seyed Al-Shohada Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Cerchietti LC, Navigante AH, Bonomi MR, Zaderajko MA, Menendez PR, Pogany CE, Roth BM. Effect of topical morphine for mucositis-associated pain following concomitant chemoradiotherapy for head and neck carcinoma. Cancer. 2002 Nov 15;95(10):2230-6. doi: 10.1002/cncr.10938. PMID 12412178
- [Background] Cerchietti L. Morphine mouthwashes for painful mucositis. Support Care Cancer. 2007 Jan;15(1):115-6; author reply 117. doi: 10.1007/s00520-006-0124-8. Epub 2006 Aug 15. No abstract available. PMID 16909245